CLINICAL TRIAL: NCT01777035
Title: Early Mobilization in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-0218
Record Dates: First submitted 2013-01-16; First posted 2013-01-28 (Estimated); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Respiratory Failure
Keywords: mechanical ventilation; physical therapy; occupational therapy; ICU acquired weakness; critical illness myopathy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early physical therapy(PT) occupational therapy (OT) (Experimental): Early PT OT assessments begin on first day of study. Therapy delivered by a team consisting of physical and occupational therapists and coordinated with daily sedative interruption
  Interventions: Other: early PT OT
- standard care (No Intervention): PT OT delivered as ordered by the primary ICU team

INTERVENTIONS:
Other: early PT OT — 1. Passive range of motion (ROM) in pts who remain unresponsive despite sedative interruption.
  2. active assisted ROM in supine position.
  3. treatment is advanced to bed mobility activities
  4. sitting balance activities followed by participation in activities of daily living (ADLs) and exercises that encourage increased independence with functional tasks.
  5. progression to transfer training, and finally pre-gait training and ambulation.
  6. progression of activities dependent on patient tolerance and stability
  7. therapy sessions continue on a daily basis throughout hospital stay until return to prior level of function or is discharged.
  Arms: Early physical therapy(PT) occupational therapy (OT)

SUMMARY:
To study all ICU patients with an independent baseline functional status , who experience a critical illness requiring intubation and mechanical ventilation evaluating long-term cognitive and executive function and long term cost effectiveness in survivors who required mechanical ventilation.

DETAILED DESCRIPTION:
Immediate mobilization of mechanically ventilated (MV) ICU patients is not part of usual care in the U.S. or internationally. Our previous work supports that early mobilization through physical and occupational therapy for ICU patients on the ventilator can help them experience less delirium, spend less time in the ICU and hospital, and become more independent when they leave. To advance our knowledge in this area, large longitudinal studies are needed to understand the long-term physical, cognitive and mental health status of survivors and to test how specific ICU therapies may affect these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and MV > 24, < 96 hours
* Baseline Barthel Index Functional Score > 70, functional at home

Exclusion Criteria:

* Rapidly changing neurological conditions (e.g. stroke)
* Cardiac arrest as cause for respiratory failure
* Elevated intracranial pressure
* Pregnancy (due to inability to provide continuous fetal monitoring)
* Terminal condition (life expectancy < 6 months)
* Traumatic brain injury, multiple limb fractures, pelvic fractures,
* Severe chronic pain syndrome on admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
presence of cognitive impairment | within the first 30 days after ICU admission
presence of cognitive impairment | up to 1 year post discharge

SECONDARY OUTCOMES:
cognitive test score | up to 1 year post discharge
  includes variables
  1. orientation
  2. attention
  3. memory
  4. reasoning
  5. executive function
institution free days | up to 1 yr post discharge
  number of days not requiring inpatient admission
Insulin Resistance | day 3 of mechanical ventilation
  Measuring insulin resistance and glycemic control in patients who are still mechanically ventilated on third day of enrollment in the study

CONTACTS AND LOCATIONS:
Overall Officials: John P Kress, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Patel BK, Wolfe KS, Patel SB, Dugan KC, Esbrook CL, Pawlik AJ, Stulberg M, Kemple C, Teele M, Zeleny E, Hedeker D, Pohlman AS, Arora VM, Hall JB, Kress JP. Effect of early mobilisation on long-term cognitive impairment in critical illness in the USA: a randomised controlled trial. Lancet Respir Med. 2023 Jun;11(6):563-572. doi: 10.1016/S2213-2600(22)00489-1. Epub 2023 Jan 21. PMID 36693400
- [Derived] Wolfe KS, Patel BK, MacKenzie EL, Giovanni SP, Pohlman AS, Churpek MM, Hall JB, Kress JP. Impact of Vasoactive Medications on ICU-Acquired Weakness in Mechanically Ventilated Patients. Chest. 2018 Oct;154(4):781-787. doi: 10.1016/j.chest.2018.07.016. Epub 2018 Sep 11. PMID 30217640